CLINICAL TRIAL: NCT05507450
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study to Evaluate the Safety and Immunogenicity of Three Different Potency Levels of V181 (Dengue Quadrivalent Vaccine rDENVΔ30 [Live, Attenuated]) in Healthy Adults
Brief Title: Safety and Immunogenicity of Three V181 Dengue Vaccine Potencies in Adults (V181-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V181-003; V181-003 (Other: MSD); 2020-004501-30 (EudraCT Number)
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Dengue Disease; Dengue Virus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- V181 High-Potency Level Group (Experimental): Participants will receive a single 0.5mL subcutaneous (SC) dose of V181 High-Potency vaccine.
  Interventions: Biological: V181 High-Potency Level
- V181 Mid-Potency Level Group (Experimental): Participants will receive a single 0.5mL SC dose of V181 Mid-Potency vaccine.
  Interventions: Biological: V181 Mid-Potency Level
- V181 Low-Potency Level Group (Experimental): Participants will receive a single 0.5mL SC dose of V181 Low-Potency vaccine.
  Interventions: Biological: V181 Low-Potency Level
- Placebo (Placebo Comparator): Participants will receive a single SC 0.5 mL dose of placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V181 High-Potency Level — 0.5 mL SC dose of V181 High-Potency vaccine
  Arms: V181 High-Potency Level Group
Biological: V181 Mid-Potency Level — 0.5 mL SC dose of V181 Mid-Potency vaccine
  Arms: V181 Mid-Potency Level Group
Biological: V181 Low-Potency Level — 0.5 mL SC dose of V181 Low-Potency vaccine
  Arms: V181 Low-Potency Level Group
Biological: Placebo — 0.5 mL SC dose of placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the dengue virus-neutralizing antibody geometric mean titers (GMTs) for each of the 4 dengue serotypes (DENV1, DENV2, DENV3, and DENV4) at Day 28 post-vaccination for participants administered the V181 Low-Potency Level vaccine versus the V181 Mid-Potency Level vaccine. This study will also evaluate the safety and tolerability of 3 different V181 potency level vaccines. The primary hypothesis of the study is that the V181 Low-Potency Level vaccine is non-inferior to the V181 Mid-Potency Level vaccine for each of the 4 dengue serotypes based on GMTs at Day 28 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Male participants are eligible to participate if they agree to the following for at least 90 days after administration of study intervention: Abstain from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause).
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is NOT women of child-bearing potential; or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), or is abstinent from heterosexual intercourse as her preferred and usual lifestyle (abstinent on a long term and persistent basis), for at least 90 days after administration of study intervention. (Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.)

Exclusion Criteria:

* Has known history of dengue or zika natural infection.
* Has an acute febrile illness (temperature ≥38.0°C [≥100.4°F] oral or equivalent) occurring within 72 hours before receipt of study vaccine or placebo.
* Has a serious or progressive disease, including but not limited to cancer; uncontrolled diabetes; severe cardiac, renal, or hepatic insufficiency; or systemic autoimmune or neurologic disorder.
* Has known or suspected impairment of immunological function, including but not limited to congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, hematologic malignancy, or treatment for autoimmune diseases.
* Has a condition in which repeated venipuncture or injections pose more than minimal risk for the participant, such as hemophilia, thrombocytopenia, other severe coagulation disorders, or significantly impaired venous access.
* Has a known hypersensitivity to any component of the study vaccine or placebo, or history of severe allergic reaction (eg, swelling of the mouth and throat, difficulty breathing, hypotension or shock) that required medical intervention.
* Has received a dose of any dengue vaccine (investigational or approved) before study entry, or plans to receive any dengue vaccine (investigational or approved) for the duration of the trial.
* Has received other licensed non-live vaccines within 14 days before receipt of study vaccine or placebo, or is scheduled to receive any licensed non-live vaccine within 28 days following receipt of study vaccine or placebo. Exception: Inactivated influenza vaccine may be administered but must be given at least 7 days before receipt of study vaccine or placebo, or at least 28 days after receipt of study vaccine or placebo.
* Has received a licensed live vaccine within 28 days before receipt of study vaccine or placebo, or is scheduled to receive any live vaccine within 28 days following receipt of study vaccine or placebo.
* Has received systemic corticosteroids (equivalent of ≥2 mg/kg/day of prednisone or ≥20 mg/d for persons weighing >10 kg) for ≥14 consecutive days and has not completed treatment at least 30 days before study entry or is expected to receive systemic corticosteroids at aforementioned dose and duration within 28 days following receipt of study vaccine or placebo. (Note: Topical and inhaled/nebulized steroids are permitted.)
* Has received systemic corticosteroids exceeding physiologic replacement doses (approximately 5 mg/day prednisone equivalent) within 14 days before vaccination.
* Has received immunosuppressive therapies, including chemotherapeutic agents used to treat cancer or other conditions, treatments associated with organ or bone marrow transplantation, or autoimmune disease, within 6 months before receipt of study vaccine or placebo, or plans to receive immunosuppressive therapies within 28 days following receipt of study vaccine or placebo.
* Has received a blood transfusion or blood products (including immunoglobulins) within 6 months before receipt of a study vaccine or placebo, or plans to receive a blood transfusion or blood products (including immunoglobulins) within 28 days following receipt of study vaccine or placebo.
* Has participated in another clinical study of an investigational product within 6 months before signing the informed consent, or plans to participate in another interventional clinical study at any time during the duration of the current clinical study. Participants enrolled in observational studies may be included; these will be reviewed on a case-by-case basis for approval by the Sponsor.
* Has planned donation of blood, eggs, or sperm at any time from signing the informed consent through 90 days post-vaccination.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1271 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (32):
- United States (6):
  - California Research Foundation ( Site 0114), San Diego, California
  - Advanced Medical Research Institute ( Site 0115), Miami, Florida
  - Rochester Clinical Research, Inc. ( Site 0122), Rochester, New York
  - University of Texas Medical Branch ( Site 0113), Galveston, Texas
  - IMA Clinical Research San Antonio ( Site 0111), San Antonio, Texas
  - Alliance for Multispecialty Research LLC (AMR - Norfolk) ( Site 0123), Norfolk, Virginia
- Australia (6):
  - Paratus Clinical Research Western Sydney ( Site 0007), Blacktown, New South Wales
  - Emeritus Research ( Site 0010), Botany, New South Wales
  - USC Clinical Trials Moreton Bay ( Site 0001), Morayfield, Queensland
  - USC Clinical Trials Sunshine Coast ( Site 0005), Sippy Downs, Queensland
  - USC Clinical Trials Brisbane (South Bank) ( Site 0006), South Brisbane, Queensland
  - Emeritus Research ( Site 0009), Camberwell, Victoria
- Canada (4):
  - Diex Recherche Quebec Inc. ( Site 0022), Québec, Quebec
  - Diex Recherche Joliette ( Site 0023), Saint-Charles-Borromée, Quebec
  - Diex Recherche Sherbrooke Inc. ( Site 0024), Sherbrooke, Quebec
  - Diex Recherche Victoriavile Inc. ( Site 0021), Victoriaville, Quebec
- Finland (9):
  - FVR, Kokkolan rokotetutkimusklinikka ( Site 0037), Kokkola, Keski-Pohjanmaa
  - FVR, Oulun rokotetutkimusklinikka ( Site 0032), Oulu, North Ostrobothnia
  - FVR, Tampereen rokotetutkimusklinikka ( Site 0039), Tampere, Pirkanmaa
  - FVR, Porin rokotetutkimusklinikka ( Site 0033), Pori, Satakunta
  - FVR, Seinäjoen rokotetutkimusklinikka ( Site 0040), Seinäjoki, South Ostrobothnia
  - FVR, Turun rokotetutkimusklinikka ( Site 0031), Turku, Southwest Finland
  - FVR, Espoon rokotetutkimusklinikka ( Site 0036), Espoo, Uusimaa
  - FVR, Etelä-Helsingin rokotetutkimusklinikka ( Site 0038), Helsinki, Uusimaa
  - FVR, Itä-Helsingin rokotetutkimusklinikka ( Site 0035), Helsinki, Uusimaa
- Germany (3):
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen-Division of Infectious Diseases and Tropical (, München, Bavaria
  - Berliner Centrum für Reise- und Tropenmedizin ( Site 0043), Berlin
  - Bernhard Nocht Institute for Tropical Medicine ( Site 0041), Hamburg
- Israel (3):
  - Rambam Health Care Campus-Oncology ( Site 0053), Haifa
  - Hadassah Medical Center-Clinical Reaserch Unit ( Site 0052), Jerusalem
  - Sheba Medical Center-Early Phase Clinical Trials Unit ( Site 0051), Ramat Gan
- Kaohsiung Medical University Hospital-Infectious diseases Division, Department of Internal Medicine, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult males or females, in generally good health, between 18 to 50 years of age, and without a history of dengue or Zika natural infection or prior receipt of any other dengue vaccine were enrolled in this study.
Groups:
- V181 High-Potency Level Group: Participants received a single 0.5 mL subcutaneous (SC) dose of V181 High-Potency vaccine.
- V181 Mid-Potency Level Group: Participants received a single 0.5 mL SC dose of V181 Mid-Potency vaccine.
- V181 Low-Potency Level Group: Participants received a single 0.5 mL SC dose of V181 Low-Potency vaccine.
- Placebo: Participants received a single SC 0.5 mL dose of placebo.
Period: Overall Study
Arm/Group | V181 High-Potency Level Group | V181 Mid-Potency Level Group | V181 Low-Potency Level Group | Placebo
Started (Randomized) | 231 | 463 | 461 | 116
Vaccinated at Baseline | 231 | 461 | 459 | 115
Completed | 205 | 430 | 431 | 106
Not Completed | 26 | 33 | 30 | 10
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 22 | 20 | 20 | 7
Not completed — Randomized By Mistake Without Study Treatment | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 11 | 7 | 3
Not completed — Participant left the country | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- V181 High-Potency Level Group: Participants received a single 0.5 mL SC dose of V181 High-Potency vaccine.
- Total: Total of all reporting groups
Arm/Group | V181 High-Potency Level Group | V181 Mid-Potency Level Group | V181 Low-Potency Level Group | Placebo | Total
Number analyzed (Participants) | 231 | 463 | 461 | 116 | 1271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (9.5) | 33.1 (9.8) | 33.3 (9.3) | 33.2 (9.1) | 33.3 (9.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 129 | 265 | 262 | 59 | 715
  Male | 102 | 198 | 198 | 57 | 555
  Undifferentiated | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 51 | 55 | 20 | 157
  Not Hispanic or Latino | 195 | 396 | 389 | 94 | 1074
  Unknown or Not Reported | 5 | 16 | 17 | 2 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 0 | 3
  Asian | 15 | 32 | 33 | 6 | 86
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 2 | 0 | 6
  Black or African American | 5 | 12 | 14 | 9 | 40
  White | 207 | 406 | 400 | 100 | 1113
  More than one race | 2 | 10 | 10 | 1 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dengue Virus-Neutralizing Antibody Titers, as Measured by Virus Reduction Neutralization Test (VRNT)
Description: A dengue VRNT was conducted to assess neutralizing antibody Geometric Mean Titers (GMTs) for each of the 4 dengue vaccine serotypes (DENV1, DENV2, DENV3, and DENV4) in specimens collected from participants on Day 28 post-vaccination.
Time Frame: Day 28 post-vaccination
Population: The population analyzed was all randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses. These deviations include participant was seropositive at baseline as assessed by VRNT and missing serology results.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V181 High-Potency Level Group | V181 Mid-Potency Level Group | V181 Low-Potency Level Group | Placebo
Number analyzed (Participants) | 178 | 377 | 380 | 99
Titer
  DENV1 Serotype | 326.31 [256.52 to 415.08] | 261.10 [220.90 to 308.61] | 184.85 [153.89 to 222.03] | 10.33 [8.79 to 12.14]
  DENV2 Serotype | 815.79 [674.69 to 986.40] | 766.98 [683.66 to 860.45] | 854.59 [755.07 to 967.22] | 7.50 [7.50 to 7.50]
  DENV3 Serotype | 203.04 [162.87 to 253.12] | 135.19 [115.70 to 157.97] | 94.69 [78.92 to 113.61] | 7.20 [6.11 to 8.48]
  DENV4 Serotype | 102.13 [77.08 to 135.33] | 68.33 [55.80 to 83.67] | 64.43 [52.42 to 79.19] | 6.50 [6.50 to 6.50]

2. Primary Outcome: Percentage of Participants With Vaccine-Related Serious Adverse Events (SAEs)
Description: An SAE is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine will be determined by the investigator.
Time Frame: Up to 28 days post-vaccination
Population: The population analyzed was all randomized participants who received at least 1 dose of study intervention according to the study intervention they received.
Measure: Number; unit: Percentage of participants
Arm/Group | V181 High-Potency Level Group | V181 Mid-Potency Level Group | V181 Low-Potency Level Group | Placebo
Number analyzed (Participants) | 231 | 461 | 459 | 115
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs include pain, erythema (redness), and swelling.
Time Frame: Up to 5 days post-vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | V181 High-Potency Level Group | V181 Mid-Potency Level Group | V181 Low-Potency Level Group | Placebo
Number analyzed (Participants) | 231 | 461 | 459 | 115
Percentage of participants
  Injection site erythema | 35.5 | 21.7 | 15.0 | 1.7
  Injection site pain | 34.2 | 19.7 | 13.5 | 14.8
  Injection site swelling | 10.0 | 5.4 | 2.4 | 2.6

4. Secondary Outcome: Percentage of Participants With Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs include rash, headache, fatigue (tiredness), pyrexia (oral temperature ≥100.4 °F or 38.0 °C), myalgia (muscle pain), and arthralgia (joint pain).
Time Frame: Up to 28 days post-vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | V181 High-Potency Level Group | V181 Mid-Potency Level Group | V181 Low-Potency Level Group | Placebo
Number analyzed (Participants) | 231 | 461 | 459 | 115
Percentage of participants
  Fatigue | 52.8 | 48.6 | 44.0 | 33.9
  Pyrexia | 10.8 | 7.6 | 5.7 | 0.9
  Arthralgia | 21.2 | 12.6 | 13.1 | 7.8
  Myalgia | 32.0 | 26.5 | 24.0 | 18.3
  Headache | 54.5 | 49.9 | 46.2 | 47.0
  Rash | 55.8 | 64.0 | 68.6 | 8.7

ADVERSE EVENTS:
Time Frame: All-cause Mortality: Randomization up to 12 months post-vaccination; Serious Adverse Events: Vaccination up to 12 months post-vaccination; Non-Serious Adverse Events: Vaccination up to 28 Days post-vaccination
Description: All-cause Mortality: randomized participants; Adverse Events: randomized participants who received at least 1 dose of study intervention according to the study intervention they received
Groups:
- V181 High-Potency Level: Participants received a single 0.5 mL SC dose of V181 High-Potency vaccine.
- V181 Mid-Potency Level: Participants received a single 0.5 mL SC dose of V181 Mid-Potency vaccine.
- V181 Low-Potency Level: Participants received a single 0.5 mL SC dose of V181 Low-Potency vaccine.
- Placebo: Participants received a single 0.5 mL SC dose of placebo
Arm/Group | V181 High-Potency Level | V181 Mid-Potency Level | V181 Low-Potency Level | Placebo
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/463 | 1/461 | 0/116
Serious Adverse Events (participants affected / at risk) | 8/231 | 9/461 | 12/459 | 6/115
Other Adverse Events (participants affected / at risk) | 200/231 | 402/461 | 406/459 | 79/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V181 High-Potency Level (N=231) | V181 Mid-Potency Level (N=461) | V181 Low-Potency Level (N=459) | Placebo (N=115)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Buttock injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Self-destructive behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V181 High-Potency Level (N=231) | V181 Mid-Potency Level (N=461) | V181 Low-Potency Level (N=459) | Placebo (N=115)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 12 (13) | 24 (24) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (15) | 9 (12) | 15 (15) | 3 (3)
Fatigue (General disorders) | 122 (125) | 224 (231) | 202 (212) | 39 (43)
Injection site erythema (General disorders) | 85 (89) | 107 (108) | 76 (76) | 2 (2)
Injection site pain (General disorders) | 80 (80) | 91 (92) | 69 (69) | 18 (18)
Injection site swelling (General disorders) | 23 (23) | 25 (25) | 12 (12) | 3 (3)
Pyrexia (General disorders) | 25 (25) | 35 (35) | 26 (26) | 1 (1)
Nasopharyngitis (Infections and infestations) | 12 (12) | 31 (31) | 15 (15) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (50) | 58 (58) | 60 (60) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 74 (75) | 122 (125) | 110 (112) | 21 (21)
Headache (Nervous system disorders) | 126 (131) | 230 (240) | 212 (230) | 54 (56)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 26 (26) | 25 (26) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 129 (131) | 295 (295) | 315 (315) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT05507450/Prot_SAP_000.pdf